CLINICAL TRIAL: NCT00834626
Title: Interventional Study of Effects of Ileal Interposition With Sleeve Gastrectomy for Control of Type 2 Diabetes
Brief Title: Ileal Interposition With Sleeve Gastrectomy for Control of Diabetes
Acronym: IISG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirloskar Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KH-001
Record Dates: First submitted 2009-02-01; First posted 2009-02-03 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-08

CONDITIONS: Diabetes
Keywords: Ileal Interposition; Sleeve Gastrectomy; Type-2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgery group (Other): Interventional study of the effects of a novel metabolic procedure of Ileal Interposition with Sleeve Gastrectomy
  Interventions: Procedure: Ileal Interposition with Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Ileal Interposition with Sleeve Gastrectomy — Transposition of a segment of Ileum proximally coupled with limited /complete sleeve gastrectomy.
  Other Names: Laparoscopic Ileal Interposition surgery

SUMMARY:
Ileal interposition shifts a segment of ileum proximally to achieve maximal meal stimulated Glucagon-Like Peptide-1 secretion and coupled with a limited/complete sleeve gastrectomy (depending on the Body Mass Index), for Ghrelin reduction, helps in achieving good glycemic control in Type 2 Diabetes patients.

DETAILED DESCRIPTION:
Laparoscopically, using 6 ports, the ileum is tarnsected at 30 cms proximal to ileo-caecal junction and at 200 cms proximal to Ileo-Caecal junction;this ileal segment of 170 cms is interposed into proximal jejunum between 20-50 cms distal to Ligament of Treitz. Endo-GIA staplers and hand-sown closure was used for the 3 anastomoses. The mesenteric gaps defects were closed with 3/0 prolene sutures. Sleeve gastrectomy was done starting from antrum/body upto angle of His with a sizing bougie ranging from size 32--58 Fr.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes (as defined by American Diabetes Association criteria)of more than 1 year duration
* Body Mass Index 21 - 55 kg/m^2
* Poor glycemic control (HbA1c > 8%) despite maximal use of Oral Hypoglycemic Agents and Insulin; or good control(lower HbA1c) but requiring progressively higher drug doses.
* Gives Informed Consent for the surgery
* Postmeal C peptide > 1.0 ng/mL
* Age 25 - 75 years
* Stable weight for more than 3 months

Exclusion Criteria:

* Type 1 Diabetes
* Postmeal C peptide < 1 ng/mL
* Pregnancy
* Significant nephropathy requiring dialysis
* Coexisting systemic disease
* Previous gastric or intestinal resection surgery
* Obesity due to organic illness

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Surendra Ugale, MS, Principal Investigator — Kirloskar Hospital, Hyderabad
Locations (1):
- Kirloskar Hospital, Hyderabad, Andhra Pradesh, India

REFERENCES:
- [Background] Kumar KV, Ugale S, Gupta N, Naik V, Kumar P, Bhaskar P, Modi KD. Ileal interposition with sleeve gastrectomy for control of type 2 diabetes. Diabetes Technol Ther. 2009 Dec;11(12):785-9. doi: 10.1089/dia.2009.0070. PMID 20001679
- [Derived] Ugale S, Gupta N, Modi KD, Kota SK, Satwalekar V, Naik V, Swapna M, Kumar KH. Prediction of remission after metabolic surgery using a novel scoring system in type 2 diabetes - a retrospective cohort study. J Diabetes Metab Disord. 2014 Aug 22;13(1):89. doi: 10.1186/s40200-014-0089-y. eCollection 2014. PMID 25426451

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in Jan 2008, at Kirloskar Hospital. Recruitment completed in May 2010.
Groups:
- Surgery Group: Interventional study of the effects of a novel metabolic surgery with anatomical modifications, to give remission of Type-2 Diabetes
Period: Overall Study
Arm/Group | Surgery Group
Started | 30
1 Year Follow-up | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Surgery Group
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.233 (9.605)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Region of Enrollment [Number; unit: participants]
  India | 30

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants Not Requiring Insulin
Description: After this Metabolic surgery, usually no Insulin is required by patient after 1 month, and definitely not after 3 months
Time Frame: 1 year
Measure: Number; unit: Percentage of Participants
Groups:
- Percentage of Participants Not Requiring Insulin: Percentage of participants not requiring Insulin assessed at 1 year post-surgery
Arm/Group | Percentage of Participants Not Requiring Insulin
Number analyzed (Participants) | 30
Percentage of Participants | 90

2. Secondary Outcome: Percentage of Participants Showing Decrease in Requirement of Oral Anti-diabetic Agents
Description: Percentage of participants showing decrease in requirement of oral anti-diabetic agents taken earlier for treatment of Type-2 Diabetes, assessed at one year
Time Frame: one year
Measure: Number; unit: Percentage of Participants
Arm/Group | Surgery Group
Number analyzed (Participants) | 30
Percentage of Participants | 93

3. Primary Outcome: Percentage of Participants Having Remission of Type 2 Diabetes
Description: The number of patients who 1 year after surgery, have a normal glycated hemoglobin (HbA1c) less than 6.5% and all medication is stopped
Time Frame: One year
Measure: Number; unit: Percentage of Participants
Arm/Group | Surgery Group
Number analyzed (Participants) | 30
Percentage of Participants | 76.66

4. Secondary Outcome: Percentage of Participants Achieving Remission in Hypertension
Description: Percentage of participants achieving remission in hypertension, that is blood pressure less than 130/80 mm Hg without any anti-hypertensive medication
Time Frame: 1 year
Measure: Number; unit: Percentage of Participants
Arm/Group | Surgery Group
Number analyzed (Participants) | 30
Percentage of Participants | 90

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Surgery Group
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
Non-availability of hormonal tests like Glucagon-Like Peptide-1 estimation pre- & post-operative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No